CLINICAL TRIAL: NCT00282399
Title: Phase I/II Trial of Subcutaneous Decitabine Maximizing Genomic Demethylation in Patients With Myelodysplastic Syndrome.
Brief Title: A Clinical Trial of Decitabine in Patients With Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACO-019
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; MGI Pharma; Decitabine; Dacogen
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DACO-019 2mg/m^2 (Experimental): DACO-019 2mg/m^2 twice daily (BID)
  Interventions: Drug: Subcutaneous Decitabine
- DACO-019 5mg/m^2 (Experimental): DACO-019 5mg/m^2 BID
  Interventions: Drug: Subcutaneous Decitabine
- DACO-019 10mg/m^2 (Experimental): DACO-019 10mg/m^2 BID
  Interventions: Drug: Subcutaneous Decitabine

INTERVENTIONS:
Drug: Subcutaneous Decitabine

SUMMARY:
The purpose of this study was to determine which of the doses of decitabine maximizes genomic demethylation in patients with Myelodysplastic Syndrome (MDS).

DETAILED DESCRIPTION:
Phase I: The purpose of this study was to determine which of the subcutaneous doses of decitabine administered twice daily for 5 days maximizes genomic demethylation in patients with MDS

Phase II: To evaluate hematological responses at the dose selected in the Phase I portion of the study.

Note: This study was planned as Phase 1/2 study but only the Phase 1 part was conducted due to a change in product development strategy

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
2. Confirmed diagnosis of MDS or non-proliferative chronic myelomonocytic leukemia (CMML).

Exclusion Criteria:

1. Prior therapy with decitabine or azacytidine (Vidaza).
2. Experimental or standard drugs for the treatment of MDS within 28 days of the first day of study drug treatment.
3. Clinically significant anemia.
4. Prior history of malignancy other than MDS.
5. Any active infection.
6. Radiotherapy within 14 days prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Phase I: To determine which of the subcutaneous (SQ) doses of decitabine administered twice daily for 5 days maximizes genomic demethylation in patients with MDS. | Up to 8 cycles (224 days)
Phase II: To evaluate hematological response at the dose selected in the Phase I portion of the study. | Up to 12 cycles (336 days)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arizona Cancer Center, Tucson, Arizona
  - H Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Albert Einstein College of Medicine, The Bronx, New York

REFERENCES:
- See also: MGI PHARMA's official website — http://www.mgipharma.com